CLINICAL TRIAL: NCT02176850
Title: Safety, Tolerability and Efficacy of Micardis® (Telmisartan) in Patients With Essential Hypertension
Brief Title: Safety, Tolerability and Efficacy of Micardis® in Patients With Essential Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.314
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Micardis®
  Interventions: Drug: Micardis®

INTERVENTIONS:
Drug: Micardis®

SUMMARY:
This post-marketing surveillance study was designed to supplement under conditions of normal clinical practice the data on the safety, tolerability and efficacy of Micardis® collected during the clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with essential hypertension and a minimum age of 18 years

Exclusion Criteria: (Not applicable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of general practioners, cardiologists and specialist in internal medicine in non-hospital practice
Sampling Method: Non-Probability Sample
Enrollment: 19870 (Actual)
Dates: Start 1999-01; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Indicence of ulcera | Up to 6 months after start of study
Incidence of gastrointestinal (GI) bleedings | Up to 6 months after start of study

SECONDARY OUTCOMES:
Incidence of adverse events (GI-complaints inclusive) | Up to 6 months after start of study
Change from baseline in office blood pressure | Up to 6 months after start of study
Response rate | Up to 6 months after start of study
  full response: reduction of diastolic blood pressure (DBP) by >= 10 mmHg or final DBP <= 90 mmHg overall response: reduction of DBP by >= 7mmHg or final DBP <= 90 mmHg